CLINICAL TRIAL: NCT00484146
Title: Alterations of Immunologic Mediators During Severe Sepsis
Acronym: LAVISS_01
Status: Terminated | Type: Observational
Why Stopped: anticipated number of patients could not be reached
Sponsor: Klinikum St. Georg gGmbH (Other)
Collaborators: University of Halle Medical Faculty (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: ISRCTN34508816; ISRCTN34508816
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Severe Sepsis
Keywords: Sepsis; Early Stage; Immune System; Receptors; Cytokines
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood Samples, Plasma Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe sepsis induces significant changes in expression of insulin- and toll-like receptors, cytokines, markers of apoptosis, and activation of t- and b-lymphocytes.

DETAILED DESCRIPTION:
In patients at early stage of severe sepsis, we investigate the expression of pro- and anti-inflammatory cytokines, chemokines, adhesion-molecules, toll-like receptors, insulin-receptors, markers of apoptosis und of t- and b-cell-activation on a mRNA level.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 y
* agreement with study procedures
* 3 of 4 SIRS-criteria
* proven or highly suspected infection
* 2 or more sepsis-induced organ failures
* start of first sepsis-induced organ failure within the last 36 hours

Exclusion Criteria:

* non-agreement with study procedures
* signs of severe sepsis with organ failure > 36 hours
* chronic immuno-compromising diseases
* chronic therapy with anti-inflammatory drugs
* non-curable cancer
* chronic renal failure with hemodialysis
* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early stage of severe sepsis and septic shock
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
severity of sepsis | 96 hours after diagnosis of sepsis
  SOFA-Score

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Principal Investigator — Klinikum St. Georg gGmbH
Locations (1):
- Klinikum St. Georg gGmbH, Interdisciplinary Intensive Care Unit, Leipzig, Saxony, Germany